CLINICAL TRIAL: NCT07014917
Title: Randomized Phase II Study of Intermittent Versus Continuous Venetoclax Therapy With Acalabrutinib in Previously Untreated Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL/SLL) and Variants of This
Brief Title: Intermittent Versus Continuous Venetoclax With Acalabrutinib for CLL/SLL
Acronym: ESR-23-22182
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zulfa Omer (Other)
Responsible Party: Sponsor-Investigator, Zulfa Omer, Principal Investigator, University of Cincinnati
Organization: University of Cincinnati (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCCC-HEM-23-01
Record Dates: First submitted 2025-05-05; First posted 2025-06-11 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; CLL Variant
Keywords: Venetoclax; Acalabrutinib; CLL; SLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — venetoclax; acalabrutinib

STUDY DESIGN:
Intervention Model Description: Two-arm, open label Subjects will be randomized with 2:1 ratio into Arm A which will receive intermittent venetoclax (7days administration per cycle) + acalabrutinib and Arm B which will receive continuous venetoclax (28 days administrations per cycle) + acalabrutinib.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: intermittent venetoclax (Experimental): intermittent venetoclax (7days administration per cycle) + acalabrutinib
  Interventions: Drug: Venetoclax; Drug: Acalabrutinib
- Arm B: continuous venetoclax (Experimental): continuous venetoclax (28 days administrations per cycle) + acalabrutinib
  Interventions: Drug: Venetoclax; Drug: Acalabrutinib

INTERVENTIONS:
Drug: Venetoclax — intermittent venetoclax (7days administration per cycle) + acalabrutinib
  Arms: Arm A: intermittent venetoclax
Drug: Acalabrutinib — intermittent venetoclax (7days administration per cycle) + acalabrutinib
  Arms: Arm A: intermittent venetoclax
Drug: Venetoclax — continuous venetoclax (28 days administrations per cycle) + acalabrutinib
  Arms: Arm B: continuous venetoclax
Drug: Acalabrutinib — continuous venetoclax (28 days administrations per cycle) + acalabrutinib
  Arms: Arm B: continuous venetoclax

SUMMARY:
This is a randomized Phase II study of intermittent versus continuous venetoclax therapy with Acalabrutinib in previously untreated Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL/SLL)

DETAILED DESCRIPTION:
This study is a two-arm, open label, Phase II multicenter clinical trial designed to evaluate the intermittent and continuous venetoclax + acalabrutinib in 2 arms in previously untreated CLL/SLL.

Phase II trial will be in two separate arms using Simon's 2-stage design for each. Subjects will be randomized with 2:1 ratio into Arm A which will receive intermittent venetoclax (7days administration per cycle) + acalabrutinib and Arm B which will receive continuous venetoclax (28 days administrations per cycle) + acalabrutinib.

With this trial we are seeking to establish efficacy of the combination therapy in both treatment models (intermittent and continuous venetoclax) and to acquire pilot data characterizing the effectiveness of the combination in increasing the depth of response as reflected in the rate of uMRD CR. We will reject the null hypothesis for each arm separately if CR at Cycle 12 obtained in 8 patients in Arm A and 5 patients in Arm B and move forward for a larger phase 3 study.

A continuous toxicity monitoring model to monitor adverse events will be used. This model has been used successfully with phase II trials designed with the Simon 2-Stage. This methodology will allow us to monitor the cumulative number of toxic events after each patient is treated and hence to stop the study if the drug toxicities exceeded the prespecified toxicity boundary.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Chronic Lymphocytic Leukemia (CLL) or Small Lymphocytic Leukemia (SLL) as defined by the IWCLL including variation of flow cytometry, provided cytogenetic or mutational data are supportive of CLL/SLL diagnosis that requires therapy by one IWCLL criteria; and, must be previously untreated CLL/SLL.

   a. Note: Variation in flow cytometry is defined as patients who have atypical immunophenotyping for CLL (CD5 negative, CD23 negative or surface expression of CD79b that is bright) but clinically behave like CLL (leukocytosis, lymphadenopathy and splenomegaly) and have the FISH/Cytogenetics translocations (del 13q, trisomy 12, Del11q) or genomic features (XPO1, NOTCH1, SF3B1, FBXW7, MYD88, BIRC3, TRAF3, NFKBIE, SAMHD1, POT1, HIST1H1E, CHD2, ZMYM3, EGR2 and others) that are suggestive of CLL
2. Men and Women ≥18 years of age.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2 with no deterioration over the previous 2 weeks prior to baseline or day of first dosing.
4. Subjects must have adequate organ and marrow function as defined below:

   1. ANC ≥1,000/mcL, unless if neutropenia is due to extensive underlying CLL bone marrow disease then platelet threshold will be ANC ≥500/mcL unless WBC is > to 50 x 109/L. If WBC is > to 50 x 109/L there will be no lower threshold of ANC. Use of steroids for disease control is allowed.
   2. Platelets ≥30,000/mcL unless thrombocytopenia is due to extensive underlying CLL bone marrow disease platelets threshold will be ≥ 10, 000/mcl. Use of steroids for disease control is allowed.
   3. Total bilirubin ≤1.5 x ULN unless directly attributable to Gilbert's syndrome
   4. AST and ALT ≤3 × ULN
   5. Creatinine clearance (Cockcroft) ≥30 mL/min/1.73 m2 • CrCl by Cockcroft and Gault method: CrCl (mL/min) = (140 - age [years]) × weight (kg) × (F)a (72 × serum creatinine mg/dL a where F = 0.85 for females and F = 1 for males ≥ 30 mL/minute
5. Female subjects who are sexually active and can bear children must agree to use highly effective forms of contraception while on the study and for 2 days after the last dose of acalabrutinib.
6. Male subjects who are sexually active must agree to use highly effective forms of contraception with the addition of a barrier method (condom) during the study.
7. Men must agree to refrain from sperm donation during the study.
8. Willing and able to participate in all required evaluations and procedures in this study protocol, including swallowing tablets without difficulty.
9. Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (in accordance with national and local patient privacy regulations).

Exclusion Criteria:

1. Evidence of any active concurrent disease (such as severe or uncontrolled systemic diseases that, in the investigator's opinion, make it undesirable for the patient to participate in the study or that would jeopardize compliance with the protocol.
2. Patients with active Richter's transformation.
3. History of or ongoing confirmed central nervous system (CNS) lymphoma.
4. Received any investigational drug within 30 days or 5 half-lives (whichever is shorter) before first dose of study drug.
5. Major surgical procedure within 30 days before the first dose of study drug. Note: If a subject had major surgery, they must have recovered adequately from any toxicity and/or complications from the intervention before the first dose of study drug.
6. History of prior malignancy that could affect compliance with the protocol or interpretation of results in the opinion of the investigator, except for the following:

   1. Basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin, carcinoma in situ of the cervix, breast or prostate at any time prior to study that are adequately treated. Patients with cancer not requiring therapy (ex: early prostate cancer under observation, should be discussed with Study PI).
   2. Continuation of maintenance therapy in patients with adequately treated malignancy
   3. Other cancers not specified above that have been curatively treated by surgery and/or radiation therapy and/or chemotherapy from which subject is disease-free for ≥3 years without further treatment
7. Significant cardiovascular disease such as symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of Screening, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification at Screening.

   a. Note: Subjects with controlled, asymptomatic atrial fibrillation are allowed to enroll on study.
8. Patients with a condition that would preclude adequate absorption, distribution, metabolism, or excretion of study treatment. For example, refractory nausea and vomiting, inability to swallow the formulated product, or malabsorption syndrome; chronic gastrointestinal disease gastric restrictions, or bariatric surgery such as gastric bypass; partial or complete bowel obstruction, or previous significant bowel resection.
9. Received a live virus vaccination within 28 days of first dose of study drug.
10. Uncontrolled HIV infection.
11. History of or ongoing confirmed progressive multifocal leukoencephalopathy (PML).
12. Any active uncontrolled significant infection (e.g., bacterial, viral or fungal), including subjects with positive cytomegalovirus [CMV] DNA polymerase chain reaction [PCR]).
13. Serologic status reflecting active hepatitis B or C infection.

    1. Note: Subjects who are hepatitis B core antibody (anti-HBc) positive and who are hepatitis B surface antigen (HBsAg) negative will need to have a negative PCR result before randomization and must be willing to undergo DNA PCR testing during the study. Those who are HbsAg-positive or hepatitis B PCR positive will be excluded.
    2. Subjects who are hepatitis C antibody positive will need to have a negative PCR result before randomization. Those who are hepatitis C PCR positive will be excluded.
14. History of stroke or intracranial hemorrhage within 6 months before first dose of study drug.
15. Uncontrolled bleeding diathesis (e.g., hemophilia, von Willebrand disease).
16. Requires or receiving anticoagulation with warfarin or equivalent vitamin K antagonists.

    a. Note: DOAC or LMWH are not exclusionary.
17. Requires treatment with a strong cytochrome P450 3A (CYP3A) inhibitor or inducer. The use of strong CYP3A inhibitors within 1 week or strong CYP3A inducers within 3 weeks of the first dose of study drug is prohibited. Patient who have started those inhibitor or inducers with known dose outside above timeline will follow dose reduction schedule provided in the protocol and package insert of venetoclax and acalabrutinib.
18. Breastfeeding or pregnant.
19. Concurrent participation in another therapeutic clinical trial.
20. Current life-threatening illness, medical condition, or organ system dysfunction which, in the Investigator's opinion, could compromise the subject's safety or put the study at risk.
21. Requires treatment with P-glycoprotein (P-gp) inhibitor during venetoclax initiating and dose escalation phase.

    Note: After initiation of the study drug(s) once a stable dose is reached if P-gp inhibitors are required then these P-gp inhibitors will be allowed per the reduction tables within the protocol or per the study drug(s) package insert/IB.
22. Patients who are unable to receive Prevnar vaccination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-12-05 (Actual); Primary Completion 2028-06-05 (Estimated); Study Completion 2032-06-05 (Estimated)

PRIMARY OUTCOMES:
Complete Remission defined by the IWCLL 2018 criteria | Post 12 cycles of treatment (each cycle is 28 days)
  Complete Remission (CR) as defined by the IWCLL 2018 criteria after 12 cycles of treatment with acalabrutinib in combination with intermittent or continuous venetoclax in patients with untreated CLL/SLL.

SECONDARY OUTCOMES:
Circulating numbers of NK cells measured by flow cytometry | Pretreatment, Cycle1, Cycle4, Cycle6, Cycle9, Cycle12 and 3 months after completion of treatment (each cycle is 28 days)
  Circulating numbers of NK cells using flow cytometry in both treatment arms at pretreatment, C1, C4, C6, C9, C12 and 3 months after completion of treatment.
Circulating numbers of T cells measured by flow cytometry | Pretreatment, Cycle1, Cycle4, Cycle6, Cycle9, Cycle12 and 3 months after completion of treatment (each cycle is 28 days)
  Circulating numbers of T cells using flow cytometry in both treatment arms at pretreatment, C1, C4, C6, C9, C12 and 3 months after completion of treatment.
Overall Survival -defined as time from study randomization to death or last follow up | From date of patient baseline visit to death or last follow up (up to 5 years post treatment).
  Overall Survival (OS) defined as time from study randomization to death or last follow up
Progression Free Survival (PFS) defined as the time from study randomization to disease progression, death, or last follow up after treatment | From date of patient baseline visit to death or last follow up (up to 5 years post treatment).
  Progression Free Survival (PFS) defined as the time from study randomization to disease progression, death, or last follow up after treatment with acalabrutinib in combination with intermittent or continuous venetoclax in patients with untreated CLL/SLL.
uMRD Complete Remission (CR) defined by negative luekemia cell to 10-6 using NGS Clonoseq | Post 12 cycles of treatment (each cycle is 28 days)
  The rate of uMRD Complete Remission (CR) defined by negative luekemia cell to 10-6 using NGS Clonoseq from bone marrow and peripheral blood samples after 12 cycles of treatment with acalabrutinib in combination with intermittent or continuous venetoclax in patients with untreated CLL/SLL.
Rate of Tumor lysis syndrome | Cycle 4 of therapy (each cycle is 28 days); post intervention point of outpatient rapid dose escalation of venetoclax
  Tumor lysis syndrome (TLS) after outpatient rapid dose escalation of venetoclax in both treatment arms.
Response to vaccination measured by Levels of antibody titer | 3 months (+/- 1 month) from completion of all treatment.
  Levels of antibody titer in response to vaccination with Prevnar 20 at 3 months (+/- 1 month) from completion of all treatment.

OTHER OUTCOMES:
BAX clonal hematopoiesis using NGS | Cycle 12, 3 and 5 years post treatment (each cycle is 28 days)
  BAX clonal hematopoiesis using NGS at Cycle 12, 3 and 5 years post treatment
Development of Secondary cancer | 3- and 5-years post treatment
  Secondary cancer development at 3- and 5-years post treatment
Quality of life measured by EORTC QLQ-CLL17 survey | Baseline (prior to first dose), cycle 1, cycle 6, cycle 9 and end of cycle 12 (each cycle is 28 days)
  Quality of life measures in the intermittent and continuous venetoclax treatment groups at baseline (prior to first dose), cycle 1, cycle 6, cycle 9 and end of cycle 12.
Mechanism of toxicity | Baseline (pre-treatment) and at cycle 1,cycle 4, cycle 6, cycle 9, and cycle 12 (each cycle is 28 days)
  Mechanism of toxicity to this combination at baseline (pre-treatment) and at C1, 4, 6, 9, and C12
Mechanism of resistance | baseline (pre-treatment) and at Cycle1, Cycle4, Cycle6, Cycle9, and Cycle12 (each cycle is 28 days)
  Mechanism of resistance to this combination at baseline (pre-treatment) and at Cycle1, Cycle4, Cycle6, Cycle9, and Cycle12 (each cycle is 28 days)
BTK mutations development rate | every 6 months from year 2 of completion of therapy until year 5.
  BTK mutations development rate every 6 months from year 2 of completion of therapy till year 5.
Disease relapse rate | every 6 months from year 2 of completion of therapy untilyear 5.
  Disease relapse rate every 6 months from year 2 of completion of therapy till year 5.

CONTACTS AND LOCATIONS:
Overall Officials: Zulfa Omer, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided